CLINICAL TRIAL: NCT07370467
Title: TEMATIC-MR: Transcatheter Mitral and Tricuspid Interventions: a Cardiac Magnetic Resonance Study
Brief Title: Transcatheter Mitral and Tricuspid Interventions: a Cardiac Magnetic Resonance Study
Acronym: TEMATIC-MR
Status: Not yet recruiting | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Hospital Álvaro Cunqueiro (Other); Centro Hospitalar de Vila Nova de Gaia/Espinho (Other)
Responsible Party: Sponsor
Other Study IDs: L2-273
Record Dates: First submitted 2025-04-01; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-01

CONDITIONS: Mitral Insufficiency; Transcatheter Aortic Valve Replacement
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mitral and tricuspid valve disease represents an increasing challenge in the management of patients with heart failure and other cardiovascular diseases. In recent years, the introduction of transcatheter techniques for valve repair and replacement (TVI) has revolutionised the treatment of these diseases, particularly for patients at high surgical risk or who are not candidates for traditional surgery. However, although these procedures are increasingly popular, their long-term effectiveness in terms of cardiac remodelling is still not well understood.

Cardiac magnetic resonance (CMR) techniques, with their advanced capabilities to provide anatomical and functional details of the heart, offer a unique opportunity to assess ventricular remodelling and valve function before and after transcatheter interventions. The ESC guidelines on valvulopathies published in 2021 recommend the use of cardiac magnetic resonance imaging not only to quantify the extent of mitral and tricuspid regurgitation when echocardiography is inconclusive, but also as the gold standard for the assessment of left and right ventricular size and function (limited, however, to the availability of this method in the various centres). Currently, there are few systematic data evaluating the effect of these procedures on CMR-assessed cardiac anatomy and function. This study aims to fill this gap by creating a multicentre registry in which clinical and advanced imaging data, including 3D echocardiography and CMR, are collected to assess the impact of these therapies.

Analysis of data derived from advanced imaging will not only provide a better understanding of the mechanism of operation of transcatheter techniques, but will also provide important information for improving long-term patient outcomes by identifying potential predictors of treatment success or failure.

DETAILED DESCRIPTION:
Mitral and tricuspid valve disease represents an increasing challenge in the management of patients with heart failure and other cardiovascular diseases. In recent years, the introduction of transcatheter techniques for valve repair and replacement (TVI) has revolutionised the treatment of these diseases, particularly for patients at high surgical risk or who are not candidates for traditional surgery. However, although these procedures are increasingly popular, their long-term effectiveness in terms of cardiac remodelling is still not well understood.

Cardiac magnetic resonance (CMR) techniques, with their advanced capabilities to provide anatomical and functional details of the heart, offer a unique opportunity to assess ventricular remodelling and valve function before and after transcatheter interventions. The ESC guidelines on valvulopathies published in 2021 recommend the use of cardiac magnetic resonance imaging not only to quantify the extent of mitral and tricuspid regurgitation when echocardiography is inconclusive, but also as the gold standard for the assessment of left and right ventricular size and function (limited, however, to the availability of this method in the various centres). Currently, there are few systematic data evaluating the effect of these procedures on CMR-assessed cardiac anatomy and function. This study aims to fill this gap by creating a multicentre registry in which clinical and advanced imaging data, including 3D echocardiography and CMR, are collected to assess the impact of these therapies.

Analysis of data derived from advanced imaging will not only provide a better understanding of the mechanism of operation of transcatheter techniques, but will also provide important information for improving long-term patient outcomes by identifying potential predictors of treatment success or failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 anni
* Signing informed consent
* Patients who are candidates for transcatheter mitral or tricuspid surgery (TEER, TTVR).

Exclusion Criteria:

* Age < 18 years
* Contraindications to CMR or administration of contrast medium (gadolinium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who are candidates for transcatheter treatment of severe mitral or tricuspid insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac Remodelling | 12 months
  Assessing the impact of mitral and tricuspid transcatheter procedures on cardiac remodelling.

SECONDARY OUTCOMES:
Analize imaging data | 12 months
  * Compare valve regurgitation quantification by echocardiography with valve regurgitation quantification by MRI using traditional phase contrast and advanced sequences such as 4D flow.
  * Establish a correlation between structural changes observed by CMR and short- and long-term (at 6 months and 1 year) clinical outcomes.
  * Analysing imaging data to identify potential predictors of procedure success and improved cardiac function.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cardiologico Monzino, Milan, Milan, Italy